CLINICAL TRIAL: NCT00050180
Title: Influence of MDR1 Genotype on Indinavir and Saquinavir Pharmacokinetics in Healthy Volunteers
Brief Title: Influence of the MDR1 Genotype on Blood Levels of Indinavir and Saquinavir in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Scott R. Penzak, Pharm.D./NIH Clinical Center, National Institutes of Health
Purpose: Treatment
Other Study IDs: 030052; 03-CC-0052
Record Dates: First submitted 2002-11-25; First posted 2002-11-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-03

CONDITIONS: Healthy; HIV Infections
Keywords: P-Glycoprotein; Protease Inhibitor; Antiretrovirals; Cytochrome P450; Drug Transporters; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections | interventions — Midazolam; Indinavir; Saquinavir

INTERVENTIONS:
Drug: Midazolam
Drug: Indinavir
Drug: Saquinavir

SUMMARY:
This study will examine whether a particular type of gene (MDR1) in the body can affect blood levels of two protease inhibitors, indinavir and saquinavir, which are used to treat people with HIV. If blood levels of these drugs are too low or too high, they may not work well or may cause side effects in patients. This study will determine how MDR1 genes might affect absorption of these medicines.

Healthy normal volunteers between 18 and 50 years of age may be eligible for this study. Candidates will be screened with a medical history and blood and urine tests. The blood will be tested for:

* Routine laboratory values for assessing general health
* HIV
* MDR1 gene type
* Amount of P-glycoprotein (a protein made by the MDR1 gene) on T cells.

Participants will have blood drawn three more times, as follows:

* After one dose of the sedative midazolam (Versed(Registered Trademark)): Participants will take an 8-milligram dose of midazolam syrup by mouth. Four hours later, a single blood sample will be drawn through a needle in an arm vein. This part of the study will assess the efficiency of a certain enzyme involved in metabolizing (breaking down) indinavir and saquinavir.
* After four doses of indinavir: About a week after taking the midazolam, participants will take 800 mg of indinavir (two capsules) 3 times a day (every 8 hours) for 1 day. The following morning they will come to the clinic, where a catheter (flexible plastic tube) will be placed in an arm vein for repeated blood draws. A blood sample will be drawn, and a fourth and final dose of indinavir will be given. Seven blood samples of about a teaspoon each will then be collected through the catheter over an 8-hour period to measure blood levels of the drug.
* After 10 doses of saquinavir: About a week after the last dose of indinavir, participants will start taking 1,200 mg (6 capsules) of saquinavir soft-gelatin capsules 3 times a day for 3 days. On the fourth day, participants will come to the clinic. A catheter will be inserted into an arm vein and about 4 teaspoons of blood will be collected for routine laboratory tests and to measure saquinavir levels. A urine sample will also be collected for routine tests. Participants will then receive the tenth and final dose of saquinavir, and eight blood samples of about a teaspoon each will be collected through the catheter over an 8-hour period.

DETAILED DESCRIPTION:
The expression of P-glycoprotein, a transporter protein present in enterocytes as well as other cells involved in the absorption and distribution of HIV protease inhibitors, has been linked to a single nucleotide polymorphism (SNP) in exon 26 of the MDR1 gene, C3435T. Individuals homozygous for the T allele have reduced P-gp expression compared to CC individuals. Preliminary studies by other investigators to determine the influence of MDR1 genotype on HIV protease inhibitor pharmacokinetics have yielded inconclusive results. The primary purpose of this study is to determine the relationship, if any, between MDR1 genotypes and plasma concentrations of the HIV protease inhibitors indinavir and saquinavir. Secondary objectives of this investigation will (1) assess the relationship between CYP3A4 activity and indinavir and saquinavir exposure and (2) characterize the relationship, if any, between P-gp expression on lymphocyte surfaces and MDR1 genotype. Up to 150 subjects will be screened to enroll a total of 63 healthy volunteers (21 subjects each in the CC, TT, and CT groups). Each subject will have blood drawn for P-gp expression analysis and MDR1 genotyping at screening. Next, subjects will receive oral midazolam 8 mg for CYP3A4 phenotyping; a single blood sample will be collected 4 hours after midazolam administration for determination of midazolam and 1-hydroxymidazolam. Between 7 and 28 days after midazolam administration, subjects will receive indinavir 800 mg every 8 hours for one day and a single 800 mg dose the next morning (dose #4). Between 7 and 28 days after indinavir administration, subjects will receive saquinavir soft-gel capsules 1200 mg three times daily for 3 days and a single dose on the morning of day 4 (dose # 10). Post-dose blood samples will be collected over 8 hours following dose #4 of indinavir and dose #10 of saquinavir. Indinavir and saquinavir pharmacokinetic parameters (primarily AUC and Cmax) will be compared across MDR1 genotype groups using ANOVA with post-hoc testing. 1-hydroxymidazolam: midazolam ratios will be correlated to indinavir and saquinavir AUCs as well as compared across MDR1 genotype groups. P-gp expression on lymphocyte surfaces will be determined by flow cytometry, quantified, and compared across MDR1 genotype groups. Data from this investigation will determine whether MDR1 genotype influences protease inhibitor plasma concentrations.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females between the ages of 18 and 60 years.
  2. Healthy by medical history and physical exam
  3. Laboratory values within established guidelines for participation in clinical studies: AST less than or equal to 2 times ULN (upper limit of normal); Serum creatinine less than or equal to ULN; hemoglobin greater than or equal to 11 g/dL.
  4. Ability to abstain from ingesting grapefruit or grapefruit juice 72 hours prior to, and the days of midazolam phenotyping and indinavir and saquinavir administration.
  5. Negative serum pregnancy test for females of child-bearing potential.
  6. Females of child-bearing potential are able and willing to practice abstinence or use other effective methods of birth control during Phase II of study that do not include oral contraceptives.

EXCLUSION CRITERIA:

1. Concomitant routine therapy with any prescription, over the counter, herbal, or holistic medications, including oral contraceptives for 30 days prior to study participation.

   * Subjects must be off oral contraceptives for at least 30 days prior to blood collection for P-gp expression analysis; they must also be off oral contraceptives for at least 30 days prior to midazolam phenotyping, and indinavir and saquinavir administration.
   * Intermittent (PRN) use of acetaminophen and non-steroidal anti-inflammatory medications (i.e. ibuprofen) will be allowed during the study; these medications should not be taken prior to, or within 4 hours of midazolam administration on Day 0. These medications should not be taken during indinavir and saquinavir administration until all blood samples for pharmacokinetic analyses of the respective drugs have been obtained.
   * Subjects will be allowed to take a multivitamin with minerals, or equivalent, once daily if they desire to do so.
2. Inability to obtain venous access for sample collection.
3. Presence of Diabetes mellitus, Human immunodeficiency virus (HIV) infection, cardiac disease (hypertension; congestive heart failure etc.), renal disease (chronic or acute renal failure or insufficiency), respiratory disease (asthma requiring chronic treatment; chronic obstructive pulmonary disease) or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.
4. Positive pregnancy test or breastfeeding female.
5. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
6. Drug or alcohol use that may impair safety or adherence.
7. History of intolerance or allergic reaction (rash; hives; swollen lips; difficulty breathing) to indinavir, saquinavir or midazolam.
8. Inability or unwillingness of females of child-bearing potential, to use a non-hormonal (barrier) method of contraception throughout the study (e.g. condom diaphragm etc.).
9. Current cigarette smoker or regular smoker within the past 6 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2002-11-22; Primary Completion 2007-08-24 (Actual); Study Completion 2007-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hammer SM, Squires KE, Hughes MD, Grimes JM, Demeter LM, Currier JS, Eron JJ Jr, Feinberg JE, Balfour HH Jr, Deyton LR, Chodakewitz JA, Fischl MA. A controlled trial of two nucleoside analogues plus indinavir in persons with human immunodeficiency virus infection and CD4 cell counts of 200 per cubic millimeter or less. AIDS Clinical Trials Group 320 Study Team. N Engl J Med. 1997 Sep 11;337(11):725-33. doi: 10.1056/NEJM199709113371101. PMID 9287227
- [Background] Acosta EP, Henry K, Baken L, Page LM, Fletcher CV. Indinavir concentrations and antiviral effect. Pharmacotherapy. 1999 Jun;19(6):708-12. doi: 10.1592/phco.19.9.708.31544. PMID 10391416
- [Background] Matheny CJ, Lamb MW, Brouwer KR, Pollack GM. Pharmacokinetic and pharmacodynamic implications of P-glycoprotein modulation. Pharmacotherapy. 2001 Jul;21(7):778-96. doi: 10.1592/phco.21.9.778.34558. PMID 11444575